CLINICAL TRIAL: NCT04065906
Title: Near-infrared Spectroscopy Neurofeedback as a Treatment for Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Wu Wenjun-1, Department of Psychiatry, Xijing Hospital, The Air Force Medical University, Xijing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192044-F-1
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Neurofeedback; Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: NIRS; fNIRS; neurofeedback; attention deficit hyperactivity disorder (ADHD); children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NIRS group (Experimental): Children with ADHD, 12 sessions of NIRS feedback, for two sessions per week.
  Interventions: Behavioral: NIRS neurofeedback
- Drug group (Other): Children with ADHD, 6 weeks' treatment of either methylphenidate or tomoxetine
  Interventions: Drug: Methylphenidate or Tomoxetine
- Control group (Other): Healthy children, 12 sessions of NIRS feedback, for two sessions per week.
  Interventions: Behavioral: NIRS neurofeedback

INTERVENTIONS:
Behavioral: NIRS neurofeedback — Neurofeedback as a treatment for ADHD can be interpreted as a way to increase behavioral inhibition. A method to assess brain activity is functional near-infrared spectroscopy (NIRS), measuring hemodynamic correlates of neural activity.
  Arms: Control group; NIRS group
Drug: Methylphenidate or Tomoxetine — Methylphenidate is the first line drug of ADHD Tomoxetine is the second line drug of ADHD
  Arms: Drug group

SUMMARY:
To observe the clinical efficacy and mechanism of functional near-infrared spectroscopy imaging neurofeedback therapy for attention deficit and hyperactivity disorder.

DETAILED DESCRIPTION:
In this study, a parallel controlled study will be conducted to recruit 60 patients with ADHD, 30 patients in the fNIRS group and 30 patients in the drug group. At the same time, 30 healthy controls will be recruited. 6 weeks, 12 sessions of NIRS feedback will be given for participants in NIRS group and healthy controls. 6 weeks of first or second line medication will be given for participants of drug group. Magnetic resonance imaging will be performed at baseline for all participants. SNAP IV, PSQ, CGI will be evaluated at baseline, week 3, week 6 and week 8 for ADHD participants.

ELIGIBILITY:
For ADHD patients:

Inclusion Criteria:

* diagnosed with TD, according to the American Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5);
* aged 6-12;
* right handed;

Exclusion Criteria:

* full-scale intelligence quotient below 80(measured by Wechsler Intelligence Scale for Children，WISC)
* medical or neurological disorders, psychiatric disorders other than oppositional defiant disorder
* current participation in a psychotherapeutic treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SNAP-IV | Baseline, week 3, week 6, week 8
  Change in SNAP-IV(Swanson, Nolan, and Pelham-IV rating scales) score between groups over time

SECONDARY OUTCOMES:
Change in CGI | Baseline, week 3, week 6, week 8
  Change in CGI (Clinical Global Impression Scale) score between groups over time
Change in PSQ | Baseline, week 3, week 6, week 8
  Change in PSQ(Parent Symptom Questionnaire) score between groups over time
Change in TRS | Baseline, week 3, week 6, week 8
  Change in TRS (Conners' Teacher Rating Scale, TRS )score between groups over time

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Wu, master, Study Chair — Xijing Hospital, The Air Force Medical University; Huaning Wang, doctor, Principal Investigator — Xijing Hospital, The Air Force Medical University; Yi Zhang, professor, Principal Investigator — Xidian University
Locations (1):
- Department of Psychiatry, Xijing Hospital, The Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Inoue Y, Sakihara K, Gunji A, Ozawa H, Kimiya S, Shinoda H, Kaga M, Inagaki M. Reduced prefrontal hemodynamic response in children with ADHD during the Go/NoGo task: a NIRS study. Neuroreport. 2012 Jan 25;23(2):55-60. doi: 10.1097/WNR.0b013e32834e664c. PMID 22146580
- [Result] Mayer K, Wyckoff SN, Fallgatter AJ, Ehlis AC, Strehl U. Neurofeedback as a nonpharmacological treatment for adults with attention-deficit/hyperactivity disorder (ADHD): study protocol for a randomized controlled trial. Trials. 2015 Apr 18;16:174. doi: 10.1186/s13063-015-0683-4. PMID 25928870
- [Result] Cortese S, Ferrin M, Brandeis D, Holtmann M, Aggensteiner P, Daley D, Santosh P, Simonoff E, Stevenson J, Stringaris A, Sonuga-Barke EJ; European ADHD Guidelines Group (EAGG). Neurofeedback for Attention-Deficit/Hyperactivity Disorder: Meta-Analysis of Clinical and Neuropsychological Outcomes From Randomized Controlled Trials. J Am Acad Child Adolesc Psychiatry. 2016 Jun;55(6):444-55. doi: 10.1016/j.jaac.2016.03.007. Epub 2016 Apr 1. PMID 27238063
- [Result] Hudak J, Rosenbaum D, Barth B, Fallgatter AJ, Ehlis AC. Functionally disconnected: A look at how study design influences neurofeedback data and mechanisms in attention-deficit/hyperactivity disorder. PLoS One. 2018 Aug 10;13(8):e0200931. doi: 10.1371/journal.pone.0200931. eCollection 2018. PMID 30096196